CLINICAL TRIAL: NCT03341325
Title: Neurovascular Reactions to Animal-assisted Therapy in Patients With Severe Disorders of Consciousness (DOC): a Randomized-controlled Trial
Brief Title: Neurovascular Reactions to AAT in Patients With DOC
Acronym: AAT NIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Rehab Basel (Other); University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAT NIRS
Record Dates: First submitted 2017-10-04; First posted 2017-11-14 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-04

CONDITIONS: Consciousness Disorder; Brain Injuries
Keywords: animal-assisted therapy
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- animal-assisted intervention (Experimental): the intervention is a real animal is presented in different forms to the participants
  Interventions: Other: animal-assisted activity
- control intervention (Active Comparator): the control intervention is a stuffed toy animal is presented in different forms to the participants
  Interventions: Other: control activity

INTERVENTIONS:
Other: animal-assisted activity — a live animal (small dog and/or rabbit)
  Arms: animal-assisted intervention
Other: control activity — a stuffed toy animal
  Arms: control intervention

SUMMARY:
There is practical evidence but no scientific investigations that persons with severe disorders of consciousness can profit from animal-assisted therapy regarding their level of awareness.

The aim of this study is to investigate the effect of animal-assisted therapy on brain activity of inpatients at REHAB Basel with severe disorders of consciousness.

To do so, the frontal brain activity of 20 the inpatients at REHAB Basel in a minimally conscious state is investigated via near-infrared spectroscopy (NIRS). Moreover, 20 healthy participants are included as control subjects.

DETAILED DESCRIPTION:
Each participant will be measured in 6 sessions. Sessions take place three times a week for 2 weeks (leading up to a total of 3 experimental sessions and 3 control sessions), each lasting for about 15 minutes.

Each session consists of 5 phases, with an animal present in three of them. In the beginning, waiting (with no stimulus presented) serves as baseline measurement. Second, an animal is watched, then the animal is placed on the patient's lap and in the fourth condition, the patient can stroke the animal with the help of the present therapist. After, there is again a waiting condition.

Control sessions are comparable sessions but with a fur pet instead of a live animal as stimulus.

Measurements are: brain activity (near-infrared spectroscopy, NIRS), skin conductance (EDA), heart rate and heart rate variability assessed via photoplethysmography (PPG) during the sessions and the BAVESTA score after each session. For further behavior analysis all sessions are videotaped.

ELIGIBILITY:
Inclusion Criteria for patients:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Inpatients of REHAB Basel with severe disorder of consciousness: minimal conscious state defined via: Glasgow Coma Scale (GCS) / Coma Recovery Scale-Revised (Koma Remissions Skala, KRS/KRS-S) / BAVESTA Score
* Minimum Age of 18 years

Inclusion Criteria for healthy participants:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* History of acquired brain-injury
* Minimum age of 18 years

Exclusion Criteria:

* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* medical contraindications for contact with animals as allergy, phobia etc.
* If the patient's medication changes radically during the time of data collection (only eligible for clinical participants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Near-infrared spectroscopy (NIRS): oxygenated hemoglobin (O2HB), deoxygenated hemoglobin (HHB), total hemoglobin (HB) and blood oxygen saturation (O2Sat) | 2 weeks
  All parameters are measured in mmol/ml throughout the sessions, measured via NONIN SenSmart

SECONDARY OUTCOMES:
Galvanic Skin Response | 2 weeks
  GSR is measured throughout the sessions via ERPrec, an EEG and ERP recording Software. Skin conductance is measured in μmho.

OTHER OUTCOMES:
Heart rate / heart rate variability | 2 weeks
  Assessed via ERPrec (photoplethysmography (PPG))
Basel Vegetative State Assessment (BAVESTA) | 2 weeks
  The BAVESTA generates a score to assess function deficits in patients with severe disorders of consciousness. The scale ranges from 0 to 5 in total with a higher score indicating higher functioning in patients.
  Subscales of vegetative regulation, attention, orientation, emotional reactivity, verbal and nonverbal communication, motor activity and information processing are reported.
Behavioral coding in Noldus Observer | 2 weeks
  All sessions are videotaped and then analyzed via behavioral coding and quantified as count variables. The variables motor activity, eye gaze, emotional reactions and communication are presented as the total number of displayed behavior percentaged to the duration of a session.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hediger, Dr. phil., Principal Investigator — Swiss TPH
Locations (1):
- REHAB Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided